CLINICAL TRIAL: NCT00146094
Title: Osteopenia and Osteoporosis in HIV Infection. Prospective BMD Measurement in Antiretroviral (ARV) Treated and Untreated HIV-1 Infected Patients
Brief Title: Bone Mineral Density (BMD) in HIV Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2860
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Osteopenia; Osteoporosis
Keywords: Osteopenia; osteoporosis; bone mineral density; HIV infection; bone metabolism; Treatment Naive
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; HIV Infections | interventions — Anti-Retroviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated patient (Experimental)
  Interventions: Procedure: BMD Measurement; Drug: antiretrovirals
- Not treated patient (No Intervention)

INTERVENTIONS:
Procedure: BMD Measurement
  Arms: Treated patient
Drug: antiretrovirals — Treated with antiretrovirals
  Arms: Treated patient

SUMMARY:
Osteopenia and osteoporosis are increasingly reported in HIV-infected patients, and appear to be more frequent than in general population. However, pathogenesis remains unclear, and published studies still give non concordant results.

We therefore started a prospective study, to assess the potential role of ARV in the occurrence of osteopenia and osteoporosis. BMD evolution over a 2-years period of follow-up, will be compared between patients starting ARV therapy, and subjects without HAART (no indication of treatment). A correlation between BMD and several factors will be looked at (see below).

This study with individual direct benefice, is conducted in 3 outpatients clinics (Strasbourg, Colmar, Mulhouse) in collaboration with the rheumatologic teams. 60 patients are planned to be included over a 3-years inclusion period

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected men, Caucasian, age > 18 years, ARV-naïve

Exclusion Criteria:

* HIV-infected women, subjects < 18 years, non-Caucasian men, ARV-experienced patients, subjects not able or willing to give informed consent, endocrine disease or treatment which could affect bone metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-03 (Actual); Primary Completion 2003-03 (Actual); Study Completion 2006-12-14 (Actual)

PRIMARY OUTCOMES:
BMD evolution and modification during 2 years of follow-up, compared between treated and untreated subjects | From enrollment to the end of follow-up at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David REY, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (3):
  - Centre Hospitalier de Colmar, Colmar
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Background] Rey D, Treger M, Sibilia J, Priester M, Bernard-Henry C, Cheneau C, Javier RM. Bone mineral density changes after 2 years of ARV treatment, compared to naive HIV-1-infected patients not on HAART. Infect Dis (Lond). 2015 Feb;47(2):88-95. doi: 10.3109/00365548.2014.968610. Epub 2014 Nov 26. PMID 25426996